CLINICAL TRIAL: NCT01055626
Title: Usefulness of the Determination of Body Composition for Establishing New Cut-offs for the Diagnosis and Follow-up of Obesity and Comorbidities
Brief Title: New Body Mass Index (BMI) Cut-offs for the Diagnosis of Obesity and Comorbidities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Principal Investigator, Gema Frühbeck Martínez, MD, PhD., Clinica Universidad de Navarra, Universidad de Navarra
Other Study IDs: OBECUN-BF-01
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Obesity; Overweight; Diabetes Mellitus, Type 2
Keywords: Body mass index; Body fat; Obesity; Overweight; Diabetes Mellitus, Type 2; Air displacement plethysmography
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Obesity is a serious medical problem because it increases the risk of cardiovascular disease (CVD), type 2 diabetes mellitus, and certain forms of cancer. The definition of obesity is based on an excess of body fat, not of BMI. However, BMI is the reference used to establish a graded classification of weight relative to height. Although BMI is widely used as a simple surrogate measure of body fat and has been shown to correlate closely with adiposity, it would be more appropriate to determine body fat percentage and to use this value for classification purposes. The present study contemplates the determination of the per cent body fat with the aim of establishing new diagnostic and therapeutic criteria according to the associated comorbidities.

DETAILED DESCRIPTION:
The prevalence of overweight and obesity has increased alarmingly in the last decades. Obesity is a serious medical problem because it increases the risk of hypertension, type 2 diabetes mellitus, coronary heart disease, sleep-breathing disorders, and certain forms of cancer. Obesity is defined medically as a state of increased adipose tissue of sufficient magnitude to produce adverse health consequences. The definition of obesity is based on an excess of body fat, not of BMI. However, BMI is the reference used to establish a graded classification of weight relative to height. Although BMI is widely used as a simple surrogate measure of body fat and has been shown to correlate closely with adiposity, it would be more appropriate to determine body fat percentage and to use this value for classification purposes. The present study contemplates the determination of the per cent body fat (by air displacement plethysmography) in more than 5,000 subjects representing the whole BMI range, with the aim of establishing new diagnostic and therapeutic criteria according to the associated comorbidities. The specific objectives are: a) To know the body fat percentage means for normal weight, overweight and obesity for both sexes. b) To know the body fat percentage means for normal weight, overweight and obesity for the different age ranges. c) To analyse the relationship between body fat percentage and BMI values in order to detect misclassified individuals. d) To establish new cut-offs for body fat percentage and the normality ranges according to its relationship with cardiovascular risk factors that could be useful in the diagnosis and therapy of obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI >18.5
* No major organ disease unrelated to excess body weight

Exclusion Criteria:

* Pregnancy/lactation
* History of eating disorder or major psychiatric illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caucasian subjects able to come to Clinica Universidad de Navarra, Pamplona, Spain.
  Patients visiting the Departments of Endocrinology and Surgery of the University Clinic of Navarra for weight loss treatment as well as hospital and University staff undergoing an annual routine health check-up .
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2005-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Differences in body fat | Baseline
  For classically defined BMI categories (normalweight, overweight and obesity) body fat will be assessed by air-displacement plethysmography (Bod-Pod)

SECONDARY OUTCOMES:
Differences in glycemic control | Baseline
  For classically-defined BMI categories measurement of fasting plasma glucose, insulin HOMA as well as response to OGTT will be related to actual body adiposity.
Differences in cardiovascular risk factors | Baseline
  For classically-defined BMI categories measurement of circulating total cholesterol, LDL-cholesterol, HDL-cholesterol, fibrinogen, C-reactive protein, homocysteine, von Willebrand factor and adipokines will be related to actual body adiposity.

CONTACTS AND LOCATIONS:
Overall Officials: Gema Frühbeck, MD, PhD, Principal Investigator — Clínica Universidad de Navarra
Locations (2):
- Spain (2):
  - Clinica Universidad de Navarra - University of Navarra, Pamplona, Navarre
  - Clinica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gomez-Ambrosi J, Silva C, Galofre JC, Escalada J, Santos S, Gil MJ, Valenti V, Rotellar F, Ramirez B, Salvador J, Fruhbeck G. Body adiposity and type 2 diabetes: increased risk with a high body fat percentage even having a normal BMI. Obesity (Silver Spring). 2011 Jul;19(7):1439-44. doi: 10.1038/oby.2011.36. Epub 2011 Mar 10. PMID 21394093
- [Result] Gomez-Ambrosi J, Silva C, Galofre JC, Escalada J, Santos S, Millan D, Vila N, Ibanez P, Gil MJ, Valenti V, Rotellar F, Ramirez B, Salvador J, Fruhbeck G. Body mass index classification misses subjects with increased cardiometabolic risk factors related to elevated adiposity. Int J Obes (Lond). 2012 Feb;36(2):286-94. doi: 10.1038/ijo.2011.100. Epub 2011 May 17. PMID 21587201
- [Derived] Gomez-Ambrosi J, Gonzalez-Crespo I, Catalan V, Rodriguez A, Moncada R, Valenti V, Romero S, Ramirez B, Silva C, Gil MJ, Salvador J, Benito A, Colina I, Fruhbeck G. Clinical usefulness of abdominal bioimpedance (ViScan) in the determination of visceral fat and its application in the diagnosis and management of obesity and its comorbidities. Clin Nutr. 2018 Apr;37(2):580-589. doi: 10.1016/j.clnu.2017.01.010. Epub 2017 Jan 28. PMID 28187933
- [Derived] Gomez-Ambrosi J, Silva C, Catalan V, Rodriguez A, Galofre JC, Escalada J, Valenti V, Rotellar F, Romero S, Ramirez B, Salvador J, Fruhbeck G. Clinical usefulness of a new equation for estimating body fat. Diabetes Care. 2012 Feb;35(2):383-8. doi: 10.2337/dc11-1334. Epub 2011 Dec 16. PMID 22179957